CLINICAL TRIAL: NCT01226797
Title: A RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED PHASE 2 STUDY TO EVALUATE THE EFFICACY AND SAFETY OF ORAL PF-04136309 500 MG BID IN SUBJECTS WITH CHRONIC HCV INFECTION AND RAISED AMINOTRANSFERASES
Brief Title: Safety And Efficacy Of Oral PF-4136309 In Patients With Chronic Hepatitis C Infection And Abnormal Liver Enzymes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A9421016
Record Dates: First submitted 2010-10-21; First posted 2010-10-22 (Estimated); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2022-09

CONDITIONS: Hepatitis C, Chronic
Keywords: Chronic HCV infection; raised ALT; transaminitis; HCV infection
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — PF-04136309

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- PF-04136309 (Active Comparator)
  Interventions: Drug: PF-04136309

INTERVENTIONS:
Drug: Placebo — Take 4 capsules twice daily 12 hours apart with water. Swallow whole.
  Arms: Placebo
Drug: PF-04136309 — Take 4 capsules twice daily 12 hours apart with water. Swallow whole.
  Arms: PF-04136309

SUMMARY:
This study will evaluate the effect of PF-04136309 in patients with chronic hepatitic C virus infection and abnormal liver enzymes.

DETAILED DESCRIPTION:
Study recruitment was stopped on Dec 15, 2011 due to difficulty in enrolling the targeted number of patients. Subjects currently enrolled into the study will complete the study as per protocol. There were no safety concerns involved in the decision to stop enrollment. The new anticipated Last Subject Last Visit (LSLV) is February 2012.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HCV infection
* ALT >1.5 but <10 times upper limit of normal

Exclusion Criteria:

* Decompensated or severe liver disease defined by one or more of the following criteria:

Prior liver biopsy showing cirrhosis.

* International Normalized Ratio (INR) greater than or equal to 1.5.
* Total bilirubin greater than or equal to 1.5X ULN, or >2X ULN for unconjugated bilirubin.
* Serum albumin below normal.
* ALT or aspartate aminotransferase (AST) >10 x ULN.
* Evidence of portal hypertension including splenomegaly, ascites, encephalopathy, and/or esophageal varices.
* Presence of human immunodeficiency virus (HIV).
* Co-infection with hepatitis B virus (HBV).
* Co-infection with Epstein Barr Virus (EBV) and/or Cytomegalovirus (CMV).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-01-17 (Actual); Primary Completion 2012-02-09 (Actual); Study Completion 2012-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- Hong Kong (2):
  - The Chinese University of Hong Kong,, Prince of Wales Hospital, Shatin, New Territories,, Hong Kong
  - The University of Hong Kong,, Hong Kong
- India (3):
  - Manipal Hospital, Bangalore, Karnataka
  - Seth G. S. Medical College & King Edward Memorial Hospital,, Mumbai, Maharashtra
  - Institute of Liver & Biliary Sciences, New Delhi
- Singapore General Hospital, Singapore, Singapore
- South Korea (2):
  - Seoul National University Hospital, Department of Internal Medicine, Seoul
  - Severance Hospital, Yonsei University College of Medicine, Division of Gastroenterology, Seoul
- Taiwan (2):
  - Chung-Ho Memorial Hospital, Kaohsiung Medical University, Kaohsiung City
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9421016&StudyName=Safety%20And%20Efficacy%20Of%20Oral%20PF-4136309%20In%20Patients%20With%20Chronic%20Hepatitis%20C%20Infection%20And%20Abnormal%20Liver%20Enzymes

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-04136309: PF-04136309 administered orally as four 125 milligram (mg) capsules twice daily for up to 4 weeks.
- Placebo: PF-04136309 matched placebo capsules administered as four capsules twice daily for up to 4 weeks.
Period: Overall Study
Arm/Group | PF-04136309 | Placebo
Started | 12 | 12
Completed | 10 | 11
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — No longer willing to participate | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- PF-04136309: PF-04136309 administered orally as four 125 mg capsules twice daily for up to 4 weeks.
- Total: Total of all reporting groups
Arm/Group | PF-04136309 | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Customized [Count of Participants; unit: Participants]
  18 to 44 years | 1 | 2 | 3
  45 to 64 years | 11 | 10 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Response in Serum Alanine Aminotransferase (ALT) Level at Week 4
Description: Responder was defined as a participant who experienced reduction in ALT of greater than or equal to (>=) 30 percent (%) of the baseline value. Baseline ALT value was defined as mean of measurements collected at screening visits 1 and 2 and pre-dose Day 1. ALT levels were determined at central lab.
Time Frame: Week 4
Population: Full Analysis Set (FAS): all randomized participants who had a baseline value and at least 1 post-baseline value. Missing data was imputed using last observation carried forward (LOCF).
Measure: Number; unit: Percentage of participants
Arm/Group | PF-04136309 | Placebo
Number analyzed (Participants) | 12 | 11
Percentage of participants | 25.00 | 36.36
Statistical Analysis 1: Comparison: PF-04136309 vs Placebo; Test type: Superiority or Other; p = 0.6668, Fisher Exact; Odds Ratio (OR) = 0.5834, 95% CI 2-sided [0.10 to 3.51] — Odds-ratio and confidence interval obtained from logistic regression with treatment as fixed effect

2. Secondary Outcome: Percentage of Participants With a Response in Serum Aspartate Aminotransferase (AST) Level From Baseline at Week 4
Description: AST responder status was defined as a reduction in AST >= 30% of the baseline value and or normalization. Baseline AST level was defined as the mean of measurements collected on screening visit 1 and pre-dose Day 1. AST levels were determined at central lab.
Time Frame: Week 4
Population: FAS population included all randomized participants who had a baseline value and at least 1 post-baseline value. Missing data was imputed using LOCF.
Measure: Number; unit: Percentage of participants
Arm/Group | PF-04136309 | Placebo
Number analyzed (Participants) | 12 | 11
Percentage of participants | 8.33 | 36.36
Statistical Analysis 1: Comparison: PF-04136309 vs Placebo; Test type: Superiority or Other; p = 0.1550, Fisher Exact; Odds Ratio (OR) = 0.1591, 95% CI 2-sided [0.01 to 1.73] — Odds-ratio and confidence interval obtained from logistic regression with treatment as fixed effect

3. Secondary Outcome: Change From Baseline in Serum ALT at Weeks 1, 2, 3 and 4
Description: Baseline ALT value was defined as mean of measurements collected at screening visits 1 and 2 and pre-dose Day 1.
Time Frame: Baseline, Weeks 1, 2, 3 and 4
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: International units per liter
Arm/Group | PF-04136309 | Placebo
Number analyzed (Participants) | 12 | 11
International units per liter
  Change at Week 1 | 11.75 [-11.08 to 34.58] | -13.70 [-37.56 to 10.16]
  Change at Week 2 | -9.40 [-28.75 to 9.94] | -22.89 [-43.11 to -2.68]
  Change at Week 3 | -9.90 [-34.77 to 14.97] | -25.08 [-51.07 to 0.92]
  Change at Week 4 | -8.25 [-35.36 to 18.85] | -32.87 [-61.20 to -4.54]
Statistical Analysis 1: Comparison: PF-04136309 vs Placebo; At Week 1; Test type: Superiority or Other; p = 0.1259, ANCOVA — Treatment as fixed effect and baseline as covariate; Mean Difference (Final Values) = 25.45, 95% CI 2-sided [-7.79 to 58.69]
Statistical Analysis 2: Comparison: PF-04136309 vs Placebo; At Week 2; Test type: Superiority or Other; p = 0.3297, ANCOVA — Treatment as fixed effect and baseline as covariate; Mean Difference (Final Values) = 13.49, 95% CI 2-sided [-14.67 to 41.66]
Statistical Analysis 3: Comparison: PF-04136309 vs Placebo; At Week 3; Test type: Superiority or Other; p = 0.3925, ANCOVA — Treatment as fixed effect and baseline as covariate; Mean Difference (Final Values) = 15.17, 95% CI 2-sided [-21.04 to 51.39]
Statistical Analysis 4: Comparison: PF-04136309 vs Placebo; At Week 4; Test type: Superiority or Other; p = 0.2080, ANCOVA — Treatment as fixed effect and baseline as covariate; Mean Difference (Final Values) = 24.62, 95% CI 2-sided [-14.85 to 64.09]

4. Secondary Outcome: Serum ALT at Baseline
Description: Baseline ALT level was defined as the mean of measurements collected on Screening visits 1 and 2 and pre-dose Day 1.
Time Frame: Baseline
Population: FAS population included all randomized participants who had a baseline value and at least 1 post-baseline value; Observed data
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | PF-04136309 | Placebo
Number analyzed (Participants) | 12 | 11
International units per liter | 132.2 (61.57) | 154.7 (81.47)

5. Secondary Outcome: Change From Baseline in Serum AST at Weeks 1, 2, 3 and 4
Description: Baseline AST level was defined as the mean of measurements collected on screening visit 1 and pre-dose Day 1.
Time Frame: Baseline, Weeks 1, 2, 3 and 4
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: International units per liter
Arm/Group | PF-04136309 | Placebo
Number analyzed (Participants) | 12 | 11
International units per liter
  Change at Week 1 | 5.90 [-9.68 to 21.47] | -15.98 [-32.25 to 0.30]
  Change at Week 2 | -5.60 [-20.04 to 8.84] | -14.89 [-29.98 to 0.20]
  Change at Week 3 | -1.65 [-18.64 to 15.33] | -15.74 [-33.49 to 2.01]
  Change at Week 4 | 5.22 [-17.48 to 27.93] | -23.97 [-47.70 to -0.24]
Statistical Analysis 1: Comparison: PF-04136309 vs Placebo; At Week 1; Test type: Superiority or Other; p = 0.0577, ANCOVA — Treatment as fixed effect and baseline as covariate; Mean Difference (Final Values) = 21.87, 95% CI 2-sided [-0.78 to 44.53]
Statistical Analysis 2: Comparison: PF-04136309 vs Placebo; At Week 2; Test type: Superiority or Other; p = 0.3669, ANCOVA — Treatment as fixed effect and baseline as covariate; Mean Difference (Final Values) = 9.30, 95% CI 2-sided [-11.71 to 30.30]
Statistical Analysis 3: Comparison: PF-04136309 vs Placebo; At Week 3; Test type: Superiority or Other; p = 0.2482, ANCOVA — Treatment as fixed effect and baseline as covariate; Mean Difference (Final Values) = 14.09, 95% CI 2-sided [-10.62 to 38.80]
Statistical Analysis 4: Comparison: PF-04136309 vs Placebo; At Week 4; Test type: Superiority or Other; p = 0.0801, ANCOVA — Treatment as fixed effect and baseline as covariate; Mean Difference (Final Values) = 29.19, 95% CI 2-sided [-3.84 to 62.22]

6. Secondary Outcome: Serum AST at Baseline
Description: Baseline AST level was defined as the mean of measurements collected on screening visit 1 and pre-dose Day 1.
Time Frame: Baseline
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | PF-04136309 | Placebo
Number analyzed (Participants) | 12 | 11
International units per liter | 96.6 (47.29) | 110.6 (48.47)

7. Secondary Outcome: Change From Baseline in Methacetin Breath Test (BreathID) at Weeks 1 and 4
Description: After drinking 13ˆC-methacetin, participants breath was collected using a BreathID® collection system for approximately 60 minutes and the ratio of 13ˆCO2:12ˆCO2 were determined to monitor the function of the liver. Results to be reported in ratio.
Time Frame: Baseline, Weeks 1 and 4
Population: Data for this outcome measure was not collected because there was a change in planned analysis owing to low enrolment number in the study.
Arm/Group | PF-04136309 | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline in Enhanced Liver Fibrosis Test (ELF) at Week 4
Description: Markers of fibrosis assessed in the ELF test comprise hyaluronic acid (HA), tissue inhibitor of matrix metalloproteinase 1 (TIMP-1), and amino terminal peptide of pro-collagen III (PIIINP). The HA ranges from 0 to 1000 in ng/mL; the TIMP-1 ranges from 0 to 3000 ng/mL; and the PIIINP tissue ranges from 0 to 151 in nanograms/milliliter (ng/mL). ELF algorithm calculates a discriminant score (DS) specified by DS = -7.412 plus (+) 0.681 times (*)ln(HA)+ 0.494 * ln(TIMP1)+ 0.775 * ln(PIIINP). Results to be reported in discriminant score.
Time Frame: Baseline, Week 4
Population: as for outcome 7
Arm/Group | PF-04136309 | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-04136309
Description: Cmax was defined as maximum observed plasma concentration of PF-04136309.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8 and 12 hours post-dose on Day 28
Population: Pharmacokinetic (PK) parameter analysis set included all enrolled participants treated and who had at least 1 of the PK parameters of interest. Here, "Overall Number of Participants Analyzed" signifies number of participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | PF-04136309
Number analyzed (Participants) | 11
Nanogram per milliliter | 3448 (1098.8)

10. Secondary Outcome: Plasma Decay Half-Life (t1/2) of PF-04136309
Description: Plasma decay half-life was the time measured for the plasma concentration to decrease by one half.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8 and 12 hours post-dose on Day 28
Population: PK parameter analysis set included all enrolled participants treated and who had at least 1 of the PK parameters of interest. Here, "Overall Number of Participants Analyzed" signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | PF-04136309
Number analyzed (Participants) | 10
Hours | 14.71 (1.4594)

11. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of PF-04136309
Description: AUCtau was defined as area under the concentration curve from time zero to end of dosing interval of PF-04136309.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8 and 12 hours post-dose on Day 28
Population: as for outcome 10
Measure: Geometric Mean (Standard Deviation); unit: Nanograms*hour per milliliter
Arm/Group | PF-04136309
Number analyzed (Participants) | 10
Nanograms*hour per milliliter | 12940 (6945.8)

12. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-04136309
Description: Tmax was defined as time to reach maximum observed plasma concentration of PF-04136309.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 6, 8 and 12 hours post-dose on Day 28
Population: as for outcome 10
Measure: Median (Full Range); unit: Hours
Arm/Group | PF-04136309
Number analyzed (Participants) | 11
Hours | 0.500 [0.500 to 2.00]

13. Secondary Outcome: Change From Baseline in Phosphorylated Extracellular Signal- Regulated Kinase (p-ERK) Levels at Week 2 and 4
Description: p-ERK is a biomarker used to assess bioavailability of PF-04136309. Baseline p-ERK level defined as the last pre-dose measurement.
Time Frame: Baseline, Week 2 and 4
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of p-ERK
Arm/Group | PF-04136309 | Placebo
Number analyzed (Participants) | 12 | 11
Percentage of p-ERK
  Change at Week 2 | -19.00 [-28.54 to -9.46] | 3.06 [-6.49 to 12.60]
  Change at Week 4 | -19.39 [-25.79 to -12.99] | -3.05 [-9.74 to 3.63]
Statistical Analysis 1: Comparison: PF-04136309 vs Placebo; At Week 2; Test type: Superiority or Other; p = 0.0031, ANCOVA — Treatment as fixed effect and baseline as covariate; Mean Difference (Final Values) = -22.06, 95% CI 2-sided [-35.67 to -8.44]
Statistical Analysis 2: Comparison: PF-04136309 vs Placebo; At Week 4; Test type: Superiority or Other; p = 0.0015, ANCOVA — Treatment as fixed effect and baseline as covariate; Mean Difference (Final Values) = -16.34, 95% CI 2-sided [-25.64 to -7.04]

14. Secondary Outcome: Baseline p-ERK
Description: as for outcome 13
Time Frame: Baseline
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of p-ERK
Arm/Group | PF-04136309 | Placebo
Number analyzed (Participants) | 12 | 11
Percentage of p-ERK | 29.63 (24.451) | 23.94 (16.435)

ADVERSE EVENTS:
Description: The same event may appear as both an adverse events (AE) and a serious adverse events (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-04136309 | Placebo
Serious Adverse Events (participants affected / at risk) | 2/12 | 0/12
Other Adverse Events (participants affected / at risk) | 8/12 | 3/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04136309 (N=12) | Placebo (N=12)
Sinus bradycardia (Cardiac disorders) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04136309 (N=12) | Placebo (N=12)
Abdominal discomfort (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 6 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Hot flush (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Study recruitment stopped early due to difficulty in enrolling enough participants. Study terminated early due to a recommendation to terminate further development of PF-04136309 in this indication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.